CLINICAL TRIAL: NCT05701332
Title: Effect of Intravesical B.C.G and Gemcitabine on Semen Quality and Testicular Volume in Patients With Non-muscle Invasive Bladder Cancer Patients
Brief Title: Effect of Intravesical B.C.G and Gemcitabine on Semen Quality and Testicular Volume
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelhafeez Elsayed, Resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: local drugs on semen
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Urothelial Carcinoma Bladder; Sperm Count, Low; Testis; Fibrosis
MeSH Terms: conditions — Oligospermia; Fibrosis | interventions — BCG Vaccine; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCG (Experimental): 6 doses of intravesical BCG
  Interventions: Biological: Bacillus Calmette Guerin

INTERVENTIONS:
Biological: Bacillus Calmette Guerin — effect of local B.C.G and Gemcitabine on semen parametes and testicular volume
  Other Names: Gemcitabine

SUMMARY:
To evaluate the effects of local intravesical B.C.G and gemcitabine on semen quality and testicular volume.

DETAILED DESCRIPTION:
Local chemotherapy has become one of the alternative strategies in treatment of cancer as many side effects on organs in human body. Despite this, also local chemotherapy has adverse effects too. One of these cancers in which local chemotherapy is used and one of the most five prevalent cancers in Egyptian men and the 3rd highest incidence numbers for specific cancer cases in Egypt in 2020,also It represents the 3rd highest mortality number from cancer in Egypt by 19% of men's mortality is bladder cancer. It is divided according to the staging system into 2 main types: the non-muscle invasive (T1) and muscle invasive (T2).The most common method used to treat T1 baldder cancer are TURT followed by local intravesical immunotherapy (like Bacillus Calmette Guerin) and chemotherapy (Gemcitabine and Mitomycin C). These drugs systemically can cause side effects like urgency, frequency, low grade fever, malaise, effect on high proliferative tissues like bone marrow, skin, hair, and seminiferous tubules….etc. Some rare side effects are acute respiratory distress syndrome and hepatic toxicity. The effect of these drugs on seminiferous tubules is still a controversy as most of the research field is focusing on systemic use, also the lack of researches focusing on local intravesical use. It can cause infertility especially in young patients with cancer who seek fertility and they are not married or not having children. The problem of fertility and urogenital cancer is multifactorial and there is a gap of knowledge as low incidence number of bladder cancer in young patients and the lack of he studies focusing on fertility in cancer patients. This study is going to unmask the mystery of one of local immunotherapy and immunotherapy and there effect on semen and testicles.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients from 20 to 60's year old (the years of reproductive active men)
2. Non muscle invasive bladder (T1 or less) urothelial carcinoma who are elected to intravesical immunotherapy or chemotherapy after TURT

Exclusion Criteria:

i. T1 carcinomas of bladder in which intravesical immunotherapy and chemotherapy is contraindicated ii. Patients under conditions that may affect sperm number, e.g. Systemic chemotherapy, radiotherapy and previous history of genitourinary tuberculosis, Prostatic carcinoma,…etc iii. Abnormal semen parameters or abnormal hormonal profile (hypogonadism) that interfere with the study, especially azoospermia and aspermia

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
decrease of one or more semen parameters | after 3 month of the 1st semen analysis
  According the 6th edition of WHO criteria of semen analysis, The main outcome is any decrease of one or more semen parameters like number of sperms less than 39 million totally, decrease in normal forms less than 4%, decrease in total motility less than 40% or progressive motility less than 30%, decrease in viability less than 54%, decrease in semen volume less than 1.5 ml.

SECONDARY OUTCOMES:
testicular volume | after 3 month of the 1st scrotal Ultrasound
  change in testicular volume less than 2 SD

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Eltaher, professor, Study Director — Professor . Dr; Hosny A Behnsawy, associate professor, Study Director — Professor . Dr; Mohammed H Zarzour, lecturer, Study Director — Dr

REFERENCES:
- [Background] Garg M, Sankhwar SN, Goel A, Kumar M, Singh BP, Singh V, Dalela D, Kumar A, Paul S. Effect of intravesical immunotherapy on sperm parameters in young patients with non--muscle-invasive bladder carcinoma: prospective analysis. Clin Genitourin Cancer. 2014 Jun;12(3):e83-6. doi: 10.1016/j.clgc.2013.11.012. Epub 2013 Nov 15. PMID 24411194
- [Background] 1. Humaid O. Al-Shamsi, Ibrahim H. Abu-Gheida, Faryal Iqbal, Aydah Al-Awadhi. Cancer in the Arab World.2022.SpringerNature. ISBN : 978-981-16-7944-5
- [Background] Raviv G, Pinthus JH, Shefi S, Mor Y, Kaufman-Francis K, Levron J, Weissenberg R, Ramon J, Madgar I. Effects of intravesical chemotherapy and immunotherapy on semen analysis. Urology. 2005 Apr;65(4):765-7. doi: 10.1016/j.urology.2004.10.049. PMID 15833524
- [Background] Avellino G, Theva D, Oates RD. Common urologic diseases in older men and their treatment: how they impact fertility. Fertil Steril. 2017 Feb;107(2):305-311. doi: 10.1016/j.fertnstert.2016.12.008. Epub 2017 Jan 7. PMID 28073432
- [Background] Flaig TW, Spiess PE, Agarwal N, Bangs R, Boorjian SA, Buyyounouski MK, Chang S, Downs TM, Efstathiou JA, Friedlander T, Greenberg RE, Guru KA, Guzzo T, Herr HW, Hoffman-Censits J, Hoimes C, Inman BA, Jimbo M, Kader AK, Lele SM, Michalski J, Montgomery JS, Nandagopal L, Pagliaro LC, Pal SK, Patterson A, Plimack ER, Pohar KS, Preston MA, Sexton WJ, Siefker-Radtke AO, Tward J, Wright JL, Gurski LA, Johnson-Chilla A. Bladder Cancer, Version 3.2020, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2020 Mar;18(3):329-354. doi: 10.6004/jnccn.2020.0011. PMID 32135513
- [Background] Han MA, Maisch P, Jung JH, Hwang JE, Narayan V, Cleves A, Hwang EC, Dahm P. Intravesical gemcitabine for non-muscle invasive bladder cancer. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD009294. doi: 10.1002/14651858.CD009294.pub3. PMID 34125951
- [Background] Griswold MD. Spermatogenesis: The Commitment to Meiosis. Physiol Rev. 2016 Jan;96(1):1-17. doi: 10.1152/physrev.00013.2015. PMID 26537427
- [Background] Amann RP. The cycle of the seminiferous epithelium in humans: a need to revisit? J Androl. 2008 Sep-Oct;29(5):469-87. doi: 10.2164/jandrol.107.004655. Epub 2008 May 22. PMID 18497337
- [Background] Frick J, Kunit G, Joos H, Rovan E, Talwar GP. Effect of intratesticular administration of BCG on testicular function (preliminary report). Int Urol Nephrol. 1983;15(1):71-81. doi: 10.1007/BF02082110. PMID 6629684
- [Background] Polland A, Berookhim BM. Fertility concerns in men with genitourinary malignancies: Treatment dilemmas, fertility options, and medicolegal considerations. Urol Oncol. 2016 Sep;34(9):399-406. doi: 10.1016/j.urolonc.2016.05.007. Epub 2016 Jun 6. PMID 27283219
- [Background] Mulhall JP, Applegarth LD, Oates RD, Schlegel PN. Fertility Preservation in Male Cancer Patients: Cambridge University Press; 2013.
- [Background] Boitrelle F, Shah R, Saleh R, Henkel R, Kandil H, Chung E, Vogiatzi P, Zini A, Arafa M, Agarwal A. The Sixth Edition of the WHO Manual for Human Semen Analysis: A Critical Review and SWOT Analysis. Life (Basel). 2021 Dec 9;11(12):1368. doi: 10.3390/life11121368. PMID 34947899
- [Background] Talarczyk-Desole J, Berger A, Taszarek-Hauke G, Hauke J, Pawelczyk L, Jedrzejczak P. Manual vs. computer-assisted sperm analysis: can CASA replace manual assessment of human semen in clinical practice? Ginekol Pol. 2017;88(2):56-60. doi: 10.5603/GP.a2017.0012. PMID 28326513